CLINICAL TRIAL: NCT05459571
Title: A Phase 2 Open-Label, Multicenter Study Evaluating The Safety And Efficacy of Axicabtagene Ciloleucel Concomitant With Prophylactic Steroids In Subjects With Relapsed Or Refractory Large B-Cell Lymphoma In The Outpatient Setting
Brief Title: Study of Axicabtagene Ciloleucel Given With Steroids In Participants With Relapsed Or Refractory Large B-Cell Lymphoma
Acronym: ZUMA-24
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kite, A Gilead Company (Industry)
Responsible Party: Sponsor
Organization: Gilead Sciences (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KT-US-482-0137
Record Dates: First submitted 2022-07-13; First posted 2022-07-15 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Relapsed or Refractory Large B-cell Lymphoma
MeSH Terms: conditions — Recurrence | interventions — axicabtagene ciloleucel; Cyclophosphamide; fludarabine; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Axicabtagene Ciloleucel (Experimental): Participant will receive lymphodepleting chemotherapy (cyclophosphamide 500 mg/m^2/day and fludarabine 30 mg/m^2/day) over 3 days (Days -5, -4, and -3) followed by prophylactic corticosteroid treatment with 10 mg dexamethasone on Day 0 (prior to axicabtagene ciloleucel), Day 1, and Day 2.
  Participant will receive axicabtagene ciloleucel consisting of a single infusion of chimeric antigen receptor (CAR)-transduced autologous T cells on Day 0 (following dexamethasone 10 mg) at a target dose of 2 x 10^6 cells/kg.
  Interventions: Biological: Axicabtagene Ciloleucel; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Dexamethasone

INTERVENTIONS:
Biological: Axicabtagene Ciloleucel — Administered intravenously
  Other Names: Yescarta®
Drug: Cyclophosphamide — Administered intravenously
Drug: Fludarabine — Administered intravenously
Drug: Dexamethasone — Administered orally or intravenously

SUMMARY:
The goal of this clinical study is to learn more about the study drug, axicabtagene ciloleucel, in participants with relapsed or refractory large B-cell lymphoma (LBCL) in the outpatient setting.

DETAILED DESCRIPTION:
Participants who complete at minimum 24 months follow up will be transitioned to a separate long-term follow-up study (study KT-US-982-5968) to complete the remainder of the 15-year follow-up assessments.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed large B-cell lymphoma (LBCL), including the following types defined by World Health Organization (WHO) 2016 classification, by local pathology laboratory assessment, are eligible as defined below:

  * Diffuse large B-cell lymphoma (DLBCL) not otherwise specified.
  * High-grade B-cell lymphoma (HGBL) with or without MYC and BCL2 and/or BCL6 rearrangement.
  * DLBCL associated with chronic inflammation; Epstein-Barr virus (EBV) + DLBCL.
  * Primary mediastinal (thymic) LBCL.
  * Primary cutaneous DLBCL, leg type.
  * Transformation of follicular lymphoma to DLBCL will also be included.
* Relapsed or refractory disease after 1 or more lines of therapy.
* Individuals must have received adequate prior therapy including:

  * Anti-CD20 monoclonal antibody AND
  * An anthracycline-containing chemotherapy regimen.
* At least 1 measurable lesion according to the Lugano Response Criteria for Malignant Lymphoma. Lesions that have been previously irradiated will be considered measurable only if progression has been documented following completion of radiation therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Individual agrees to outpatient treatment setting and to adhere to the prespecified clinical monitoring requirements.

Key Exclusion Criteria:

* History of autologous or allogeneic stem cell transplant.
* Prior cluster of differentiation (CD)19 targeted therapy.
* Prior chimeric antigen receptor therapy or other genetically modified T-cell therapy.
* Presence of fungal, bacterial, viral, or other infection that is uncontrolled or requiring intravenous (IV) antimicrobials for management. Simple urinary tract infection and uncomplicated bacterial pharyngitis are permitted if responding to active treatment and after consultation with the Kite medical monitor.
* Individuals with detectable cerebrospinal fluid malignant cells, brain metastases, or with a history of central nervous system (CNS) lymphoma or primary CNS lymphoma. DLBCL epidural involvement should be considered as positive CNS disease.
* In the investigator's judgment, the individual is unlikely to complete all protocol-required study visits or procedures, including follow-up visits, or comply with the study requirements for participation.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2025-11-24 (Actual); Study Completion 2025-11-24 (Actual)

PRIMARY OUTCOMES:
Percentage and Severity of Participants with Treatment-emergent Cytokine Release Syndrome (CRS) and Neurologic Events | Up to 24 months

SECONDARY OUTCOMES:
Time to Onset of CRS and Neurologic Events Following Axicabtagene Ciloleucel Administration | First infusion date of axicabtagene ciloleucel up to 24 months
Duration of CRS and Neurologic Events Following Axicabtagene Ciloleucel Administration | First infusion date of axicabtagene ciloleucel up to 24 months
Rates of Hospitalization After Axicabtagene Ciloleucel Infusion as Measured by Proportion of Hospitalized Participants Within 72 hours | First infusion date of axicabtagene ciloleucel up to 72 hours
Rates of Hospitalization After Axicabtagene Ciloleucel Infusion as Measured by Proportion of Hospitalized Participants 3 Days After Infusion Date | First infusion date of axicabtagene ciloleucel up to 3 days
Rates of Hospitalization After Axicabtagene Ciloleucel Infusion as Measured by Proportion of Hospitalized Participants Within 7 days | First infusion date of axicabtagene ciloleucel up to 7 days
Rates of Hospitalization After Axicabtagene Ciloleucel Infusion as Measured by Proportion of Hospitalized Participants Within 14 days | First infusion date of axicabtagene ciloleucel up to 14 days
Rates of Hospitalization After Axicabtagene ciloleucel Infusion as Measured by Proportion of Hospitalized Participants Within 30 days | First infusion date of axicabtagene ciloleucel up to 30 days
Duration of Initial Hospitalization After Axicabtagene Ciloleucel Infusion | First infusion date of axicabtagene ciloleucel up to 24 months
Proportion of Intensive Care Unit (ICU) Admitted Participants | Up to 24 months
Duration of ICU Admission During First Hospitalization After Axicabtagene Ciloleucel Infusion | Up to 24 months
Percentage of Participants Experiencing Treatment- Emergent Adverse Events | First infusion date of axicabtagene ciloleucel up to 24 months
Percentage of Participants Experiencing Treatment- Emergent Serious Adverse Events | First infusion date of axicabtagene ciloleucel up to 24 months
Change in the European Quality of Life Five Dimensions Five Levels Scale (EQ-5D-5L) From Baseline to Month 6 | Baseline, 6 Months
  The EQ-5D-5 levels (EQ-5D-5L) is a standardized measure of health status of the participant that provides a simple, generic measure of health for clinical and economic appraisal. EQ-5D-5L consists of 2 components: a descriptive system of the participant's health and a rating of his or her current health state on a 0-100 VAS. The descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. Rating gets recorded on a vertical VAS in which the endpoints are labeled best imaginable health state is 100 (on the top) and worst imaginable health state is 0 (on the bottom). Higher scores of EQ VAS indicate better health.
Objective Response Rate (ORR) as Assessed by Investigator Assessment | Up to 24 months
  ORR is defined as the incidence of either a complete response or a partial response by the revised international working group (IWG) response criteria for malignant lymphoma.
Complete Response (CR) Rate as Assessed by Investigator Assessment | Up to 24 months
  CR rate is defined as the incident of complete response.
Duration of response (DOR) as Assessed by Investigator Assessment | Up to 24 months
  DOR is defined as the time from first objective response to disease progression per the revised IWG response criteria for malignant lymphoma or death from any cause.
Progression-free Survival (PFS) as Assessed by Investigator Assessment | Up to 24 months
  PFS is defined as the time from the axicabtagene ciloleucel infusion date to the date of disease progression per the revised IWG response criteria for malignant lymphoma or death from any cause.
Event Free Survival (EFS) as Assessed by Investigator Assessment | Up to 24 months
  EFS is defined as the time from infusion to the earliest date of disease progression per the revised IWG response criteria for malignant lymphoma, commencement of new anti-lymphoma therapy, or death from any cause.
Overall Survival (OS) | Up to 24 months
  OS is defined as the time from axicabtagene ciloleucel infusion to the date of death.
Peak Serum Levels of Homeostatic/Proliferative Cytokines: Interleukin (IL)-2, IL-7, and IL-15 | Up to 24 months
Peak Serum Levels of Inflammatory and Immune Modulating Cytokines: IFN-γ, IL-1, IL-6, IL- 13, IL-17, IL-1, IL-1RA, Granulocyte-macrophage Colony Stimulating Factor (GM-CSF), Tumor Necrosis Factor-Alpha (TNF-α), and IL-12p40/p70 | Up to 24 months
  IFN-γ=Interferon-Gamma, IL-1RA=IL-1 Receptor Antagonist
Peak Serum Levels of Immune Effector Molecules: Granzyme A, Granzyme B, and Perforin | Up to 24 months
Peak Serum Levels of the Acute Phase Response Proteins: C-Reactive Protein (CRP), Serum Amyloid A (SAA), Soluble IL-2 Receptor Alpha (sIL-1Ra), Ferritin | Up to 24 months
Peak Serum Levels of Chemokines: IL-8, C-X-C Motif Chemokine Ligand-10 (CXCL-10), and Monocyte Chemotactic Protein-1 (MCP-1) | Up to 24 months
Blood Levels of Axicabtagene Ciloleucel Chimeric Antigen Receptor (CAR) T-cells Over Time | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Kite Study Director, Study Director — Kite, A Gilead Company
Locations (16):
- United States (16):
  - City of Hope (City of Hope National Medical Center, City of Hope Medical Center), Duarte, California
  - UCLA, Los Angeles, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - University of Maryland Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Oncology Hematology Care Clinical Trials, LLC, Cincinnati, Ohio
  - Prisma Health - Upstate, Greenville, South Carolina
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Henry-Joyce Cancer Clinic, Nashville, Tennessee
  - Methodist Healthcare System of San Antonio, San Antonio, Texas
  - Intermountain Healthcare, Murray, Utah
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gileadclinicaltrials.com/transparency-policy#Commitment
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gileadclinicaltrials.com/transparency-policy#Commitment

REFERENCES:
- [Derived] Leslie LA, Baird JH, Flinn IW, Tees M, Hoda D, Deol A, Young P, McClune B, Varadarajan I, Essell J, Fanning S, Simmons G, Clark W, Rapoport AP, Rodriguez TE, Winters JN, Davis M, Miao HM, Ray M, Fang X, Kim JJ, Oluwole OO. Outpatient axicabtagene ciloleucel for relapsed/refractory large B-cell lymphoma: ZUMA-24 primary analysis. Am J Cancer Res. 2025 Aug 15;15(8):3417-3433. doi: 10.62347/GJNN1023. eCollection 2025. PMID 40948517
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=KT-US-482-0137